CLINICAL TRIAL: NCT05145803
Title: Asymptomatic and Pre-symptomatic Transmission of SARS-CoV-2 in a Community Congregant Setting: a Study to Understand How Infection Control Practices Can Mitigate Exposure Risks
Brief Title: Asymptomatic and Pre-symptomatic Transmission of SARS-CoV-2 in a Community Congregant Setting
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Colorado School of Public Health (Other)
Collaborators: Colorado State University (Other); University of Colorado, Boulder (Other); Colorado Mesa University (Other); Regis University (Other); Denver Health Medical Center (Other); University of Colorado, Colorado Springs (Other); University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Thomas Jaenisch, Associate Professor, Colorado School of Public Health
Other Study IDs: 21-2823
Record Dates: First submitted 2021-12-01; First posted 2021-12-06 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: COVID-19; SARS-CoV2 Infection
Keywords: COVID-19 Transmission; SARS-CoV2 Transmission
MeSH Terms: conditions — COVID-19 | interventions — Diagnosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasal swabs, PVA in masks, venous blood sample [1x], dried blood spots [optional]
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- College Students: Collegiate students tested positive for SARS-CoV-2 by a molecular reference test (PCR test or antigen test) (index patients).
  Collegiate students known to be contacts of the index patients.
  Interventions: Device: Polyvinylalcohol strip [diagnostic]

INTERVENTIONS:
Device: Polyvinylalcohol strip [diagnostic] — The investigators will measure SARS-CoV-2 in exhaled breath of asymptomatic and symptomatic persons using PVA test strips embedded in face masks (FMS) - an innovative, non-invasive method for detection of SARS-CoV-2 in exhaled air. Utilizing this approach, the study aims to utilize the test results extracted from the masks to identify risk factors for SARS-CoV-2 transmission and timing of infectious period in exposed people (pre-symptomatic, asymptomatic, and symptomatic).

SUMMARY:
The overall aim of this study is to measure how transmission of COVID-19 occurs in communities - including the role of super spreaders and/or identifying conditions that may increase transmission risk, with a focus on congregant situations. In order to identify how presence of symptoms and behavior affects the transmissibility of the virus, the investigators will measure SARS-CoV-2 in exhaled breath of asymptomatic and symptomatic persons using polyvinyl alcohol (PVA) test strips embedded in face masks (Face Mask Sampling- "FMS") - an innovative, non-invasive method for detection of SARS-CoV-2 in exhaled air.

ELIGIBILITY:
Inclusion Criteria:

* Individuals age ≥ 18 years of any gender tested positive for SARS-CoV-2 by a molecular reference test (PCR test or antigen test) [INDEX PATIENTS]
* Individuals age ≥ 18 years and known to be contacts of the index patients [CONTACTS]

Exclusion Criteria:

* < age 18 years old, unable to wear a face mask due to underlying condition, not able to consent, pregnancy. In addition, signs of severe disease present at time of enrollment (e.g. difficulty breathing, pain when breathing, tightness of chest or developing irregular heart beat).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Students 18 years and older
Sampling Method: Non-Probability Sample
Enrollment: 3300 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-03-09 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
PVA strip positivity | 72 hours after sample collection

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Winstanley, PharmD, Study Director — Colorado School of Public Health; Molly Lamb, PhD, Principal Investigator — Colorado School of Public Health; May Chu, PhD, Principal Investigator — Colorado School of Public Health; Thomas Jaenisch, MD, PhD, Principal Investigator — Colorado School of Public Health
Locations (6):
- United States (6):
  - Anschutz Medical Campus, Aurora, Colorado
  - University of Colorado, Boulder, Boulder, Colorado
  - University of Colorado, Colorado Springs, Colorado Springs, Colorado
  - Denver Health, Denver, Colorado
  - Regis University, Denver, Colorado
  - Colorado State University, Fort Collins, Colorado

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jaenisch T, Lamb MM, Gallichotte EN, Adams B, Henry C, Riess J, van Sickle JT, Hawkins KL, Montague BT, Coburn C, Conners Bauer L, Kovarik J, Hernandez MT, Bronson A, Graham L, James S, Hanenberg S, Kovacs J, Spencer JS, Zabel M, Fox PD, Pluss O, Windsor W, Winstanley G, Olson D, Barer M, Berman S, Ebel G, Chu M. Investigating transmission of SARS-CoV-2 using novel face mask sampling: a protocol for an observational prospective study of index cases and their contacts in a congregate setting. BMJ Open. 2022 Nov 23;12(11):e061029. doi: 10.1136/bmjopen-2022-061029. PMID 36418127